CLINICAL TRIAL: NCT00857038
Title: Doxycycline and Airway Inflammation in COPD: A Randomised Placebo Controlled Trial Studying the Effects of Doxycycline on Airway Inflammation in Patients With Moderate and Severe Stable COPD.
Brief Title: Doxycycline and Airway Inflammation in Chronic Obstructive Pulmonary Disease (COPD)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical Center Alkmaar (Other)
Collaborators: Leiden University Medical Center (Other); University of Amsterdam (Other)
Responsible Party: Boersma, MD, PhD, Medical Center Alkmaar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M07-046
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2009-03-06 (Estimated); Status verified 2009-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Inflammation; Pulmonary Emphysema
Keywords: COPD; Inflammation; Neutrophilic; Myeloperoxidase; Doxycycline
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation; Pulmonary Emphysema | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Doxycycline 100mg daily
  Interventions: Drug: Doxycycline
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxycycline — Doxycycline tablets, 100mg daily
  Arms: 1
Drug: Placebo — Placebo tablets 100mg
  Arms: 2

SUMMARY:
COPD is a progressive pulmonary disease that is characterized by an inflammatory process in the airways and the lungs which leads to progressive airway obstruction. The inflammation is associated with tissue loss and remodelling. The investigators hypothesized that doxycycline reduces neutrophilic airway inflammation in patients with COPD. Therefore the investigators will conduct a randomized trial of doxycycline in 30 patients.

DETAILED DESCRIPTION:
Rationale:

COPD is a disease characterized by chronic inflammation and irreversible airway obstruction. Chronic inflammation lead to degradation of extracellular matrix and hereby destruction of lung parenchyma. Tetracyclines are known for their anti-inflammatory properties in diseases such as rheumatoid arthritis.

Objective:

To assess the effect of doxycycline on markers of neutrophilic inflammation and proteolytic activity in induced sputum of stable GOLD II and III COPD patients.

Study population:

Thirty patients with stable GOLD II COPD.

Intervention:

Placebo versus doxycycline in randomised design.

ELIGIBILITY:
Inclusion Criteria:

* GOLD II or III COPD (GOLD II: FEV1/FVC < 70%; 50% < FEV1 < 80% predicted, GOLD III: FEV1/FVC < 70%; 30% < FEV1 < 50% predicted ).
* Stable disease (no exacerbations in the last 3 months).
* Age > 40 yrs.
* Written informed consent.

Exclusion Criteria:

* Infections and/or use of antibiotics in the last month.
* Bacterial colonization of the airways, proven by sputum cultures or broncho-alveolar lavage (BAL).
* Allergy for tetracyclines or a history of substantial side-effects.
* Active respiratory diseases other than COPD (e.g. sarcoidosis, tuberculosis, lung cancer, bronchiectasis).
* Acute exacerbation of COPD as defined by Anthonisen et al. [10].
* Signs and/or symptoms of a current respiratory or non-respiratory infection.
* Use of oral or intravenous corticosteroids or other immunosuppressive drugs within the last month.

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-08 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
myeloperoxidase in induced sputum | 3 weeks

SECONDARY OUTCOMES:
MMP-8, MMP-9, IL-6 levels and differential cell counts in induced sputum. | 3 weeks
Lung function (FEV1) | 3 weeks
Symptom scores | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center Alkmaar, Alkmaar, North Holland, Netherlands

REFERENCES:
- [Derived] Prins HJ, Daniels JM, Lindeman JH, Lutter R, Boersma WG. Effects of doxycycline on local and systemic inflammation in stable COPD patients, a randomized clinical trial. Respir Med. 2016 Jan;110:46-52. doi: 10.1016/j.rmed.2015.10.009. Epub 2015 Oct 30. PMID 26616678